CLINICAL TRIAL: NCT04977245
Title: Mindfulness-Based Stress Reduction Intervention in Caregivers of Dementia Patients: A Randomized Clinical Trial
Brief Title: Mindfulness-Based Stress Reduction in Dementia Caregivers
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-31240
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Mindfulness Based Stress Reduction; Caregiver Burnout; Caregiver Stress Syndrome; Dementia; Dementia Frontal; Frontotemporal Dementia; Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Caregiver Burden; Dementia; Frontotemporal Dementia; Frontotemporal Lobar Degeneration | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Two groups of 20 participants. Group 1 is the control arm (online, self-guided stress reduction course) and group 2 is the intervention arm (MBSR group.)
Masking Description: Due to the nature of this study, masking is not possible. Participants and researchers must be aware of which arm they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR Intervention (Experimental): The intervention group will take part in a group-based mindfulness-based stress reduction (MBSR) program led by a certified MBSR instructor via Zoom. This MBSR program will have a shortened session length of 1.5 hours compared to the traditional 2 hours, to reduce caregiver burden. Caregivers will be trained in meditation practices, like awareness of one's breath, body scan, and loving kindness meditation. Participants will also learn about mindfulness and stress theory, and have group discussions covering topics such as self-compassion.
  Interventions: Other: Mindfulness-Based Stress Reduction
- Self-Guided Meditation eCourse (Active Comparator): Participants in the active control group will participate in a self-guided, online program named GARDEN. The self guided material teaches skills about increasing the daily experience of positive emotion as a mechanism to assist with stress coping. The program consists of eight skills introduced and discussed over an eight week period.
  Interventions: Other: Self-Guided Mindfulness eCourse

INTERVENTIONS:
Other: Mindfulness-Based Stress Reduction — Eight MBSR sessions of 1.5 hours per week
  Other Names: MBSR; Mindfulness Based Stress Reduction
  Arms: MBSR Intervention
Other: Self-Guided Mindfulness eCourse — Six weeks of a mindfulness ecourse, and two weeks of coping skills training led by a licensed neuropsychologist
  Arms: Self-Guided Meditation eCourse

SUMMARY:
Aims: The study will contribute to our understanding of how the cultivation of caregiver mindfulness might improve their overall relational well-being (Primary Outcome), their psychological well-being (Secondary Outcome), and have an impact on dementia patients' lifestyles (Other Outcome). Overall, this study will investigate the idea that the fruits of mindfulness training can be leveraged by both the caregiver and the care-recipient, improving the quality of relationship by making their interactions more mutual, connected, empathic and positive. This study aims to additionally elucidate which facets of mindfulness account for caregiver's happiness and psychological well-being.

Sample: In this study 40 dementia caregivers will be recruited to participate; 20 will be allocated to the clinical intervention group (i.e., adapted MBSR for caregivers) and 20 to the active control group. Data will be collected pre-post the start of intervention, and at a 3 month follow up.

Future orientation: This study may contribute to evidence-based knowledge concerning the efficacy of mindfulness based interventions to support caregiver empowerment, via regaining relationship satisfaction and achieving greater equanimity in the face of stressors.

DETAILED DESCRIPTION:
Caring for a family member with dementia is a very challenging task. Caregiving is associated with a hodgepodge of challenges, including negative affect, burnout, social isolation, role challenges, as well as decreased relationship quality between the caregiver and the care recipient. These conditions are often sustained over time and can implicate significant detrimental effects on the caregiver's physical and mental health, as well as their overall well-being. Criticism and emotional over-involvement expressed by the family member toward the patient seem to positively relate to the levels of caregiver strain and to reflect poor relationship quality. Mindfulness cultivates skills of non-reactivity, acceptance and awareness, which may work in the opposite direction to reactive, non-skillful coping mechanisms and seem to enhance attributes connected with individual happiness. Adopting those skills might, thus, ameliorate caregiver relationship quality and contribute in reframing the caregiving experience as more meaningful and positive.

Criticism and reactivity can be relayed by the caregiver to the patient and thus negatively affect relational well-being in the caregivers (Primary Outcome). A potential counter mechanism involves the cultivation of mindfulness skills of awareness and non-reactivity. Broadening perspective without automatically reacting may be crucial for improving the perceived relationship quality between caregiver and demented patient. Despite studies claiming a role for meditation and dispositional mindfulness in social cognition domains, there is a noteworthy gap in the literature with regard to how exactly meditation and mindfulness facets are associated with specific social cognition domains - i.e., how the focus on the experience of the present moment affects the way people perceive and interact with each other. Accordingly, very little is known about the effects of mindfulness how it may affect relationship quality in patient-caregiver couples dyads.

This study will also evaluate the effect of mindfulness skill development on the overall happiness and psychological well-being of caregivers (Secondary Outcome). Mindfulness training can help caregivers of dementia patients to be more aware of their emotional states, by enabling them to better acknowledge and accept any stressful or negative experiences they may encounter. The cultivation of self-compassion through mindfulness may help caregivers to be more kind and understanding of their role in such experiences, thus fostering self-kindness and decreasing self-judgment. These skills (acceptance, awareness, self-compassion), in turn, may lead to a decrease in rumination and allow for a newfound, more constructive appreciation of positive experiences. Caregivers of dementia patients may gain a new perspective on their role as a caregiver, potentially resulting in increased positive affect and reframe of caregiving experience as more purposeful. As an additional outcome, investigators will further explore the impact of caregiver mindfulness cultivation on the care recipient's lifestyle, manifested as frequency of engagement in specific daily activities, and the observed level of pleasure the dementia patient receives from these daily activities.

This aim of this study is to contribute to evidence-based knowledge concerning the efficacy of mindfulness-based interventions to support caregiver empowerment via improved relationship satisfaction and equanimity.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18 or older
* Caregiver for a patient with dementia in personal life and regular weekly contact with the demented patient
* English speaking
* Literate: is able to read course material
* Able to attend weekly classes online via Zoom
* Willing to be randomized and participate in one of two interventions

Exclusion Criteria:

* Are regularly practicing mindfulness meditation, mindful yoga, or similar mindfulness activities
* Currently experiencing active trauma (PTSD - unresolved, or acute stress disorder) without professional psychological assistance
* Clinical diagnosis of dementia
* Diagnosed with psychotic disorder such as schizophrenia, schizoaffective disorder or bipolar disorder according to the Diagnostic and Statistical Manual-V (DSM-V), and under antipsychotic treatment
* Undergoing treatment for substance abuse
* Vision or hearing impairments that would keep them from adequately participating in the intervention
* Any prior formal training in MBSR
* Acute suicide plans as measured by the Patient Safety Screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Experiential Avoidance in Caregiving Questionnaire (EACQ) Score | Baseline, 21 weeks
  The Experiential Avoidance in Caregiving Questionnaire (EACQ) is a 15-item self-report questionnaire measuring experiential avoidance in caregivers. Scores range 15-75, and higher scores indicate greater levels of experiential avoidance.
Change in Short Form Zarit Burden Interview (ZBI-SF) Score | Baseline, 21 weeks
  The Zarit Burden Interview (ZBI) assess the stresses experienced by caregivers of patients with dementia. The short form assesses 12 questions about the impact of the patient's disabilities on the caregiver's life, each rated from least (0) to most (4) frequent. Items are summed to calculate the ZBI total score. The ZBI total score ranges from 0 to 48; higher scores denoting more stresses experienced by caregivers.
Change in Positive Aspects of Caregiving (PAC) Scale | Baseline, 21 weeks
  The Positive Aspects of Caregiving Scale asks caregivers to rate their agreement/disagreement with 9 statements about positive aspects of caregiving on a 5-point Likert scale from "disagree a lot" to "agree a lot." Scores can range from 9 to 45 with higher scores indicating more subjective positive aspects of providing care to someone.
Change Mutuality scale of the Family Care Inventory (FCI-MS) Score | Baseline, 21 weeks
  The Mutuality Scale of the Family Care Inventory will be used for rating mutual concerns and overall relationship satisfaction. The measure consists of 15 items. Scores range from 0-60, higher scores indicate greater relationship satisfaction.
Change in Interpersonal Reactivity Index Empathic Concern (IRI-PT) Score | Baseline, 21 weeks
  The Interpersonal Reactivity Index (IRI) was designed to assess empathy, and has 28 items on a 5-point Likert scales (1 = does not describe me well to 5 = describes me very well). The perspective-taking scale assesses the extent to which individuals are able to take on others' points of view. Each of the 4 sub-scales has 7 items and scores range from 7 to 35. Higher scores indicate a greater ability to take on the perspective of other persons in social contexts.
Change in Interpersonal Reactivity Index Empathic Concern (IRI-EC) Score | Baseline, 21 weeks
  The Interpersonal Reactivity Index (IRI) was designed to assess empathy, and has 28 items on a 5-point Likert scales (1 = does not describe me well to 5 = describes me very well). The empathetic concern scale assesses the extent of individuals' concern and compassion for others. Each of the 4 sub-scales has 7 items and scores range from 7 to 35. Higher scores indicate a greater amount of empathy for others.
Change in Interpersonal Reactivity Index Personal Distress (IRI-PD) Score | Baseline, 21 weeks
  The Interpersonal Reactivity Index (IRI) was designed to assess empathy, and has 28 items on a 5-point Likert scales (1 = does not describe me well to 5 = describes me very well). The personal distress subscale assesses individuals anxiety as a result of other's negative experiences. Each of the 4 sub-scales has 7 items and scores range from 7 to 35. Higher scores indicate a greater amount of personal distress for others' negative situations.
Change in Interpersonal Reactivity Index Fantasy (IRI-FS) Score | Baseline, 21 weeks
  The Interpersonal Reactivity Index (IRI) was designed to assess empathy, and has 28 items on a 5-point Likert scales (1 = does not describe me well to 5 = describes me very well).The fantasy subscale assesses the extent to which individuals identify with fictional characters. Each of the 4 sub-scales has 7 items and scores range from 7 to 35. Higher scores indicate a greater ability to identify with fictional characters.
Change in Fears of Compassion Scale (FCS): Fear of Compassion for Others Subscale | Baseline, 21 weeks
  This scale is comprised of 10 items and assesses the compassion we feel for others, related to our sensitivity to other people's thoughts and feelings. Scores range from 0 to 40. Higher scores indicate greater fear of compassion for others.
Change in Fears of Compassion Scale (FCS): Fear of Compassion from Others Subscale | Baseline, 21 weeks
  This scale is comprised of 13 items the compassion that we experience from others and flowing into the self. Scores range from 0 to 52. Higher scores indicate greater fear of compassion from others.
Change in The Awareness of Social Inference Task SIE (TASIT-SIE) Score | Baseline, 21 weeks
  The TASIT test asks participants to watch 16 brief videos of social interactions, and answer 4 "Yes" or "No" questions per video. Answering these questions requires the ability to make inferences based on sarcasm, facial expressions, and other social elements seen in the videos, and measures socioemotional sensitivity. Higher scores indicate better ability to make real-world social inferences.
Change in Humor Picture Test Score | Baseline, 21 weeks
  The Humor Picture test presents 8 different scenarios each with 4 potentially humorous outcomes that may be correct funny, straightforward, humorous nonsequitur, or unrelated nonsequitur, and is used to measure humor comprehension. Responses to each of the 4 categories are added together to allow 0-8 points in each category.
Change in Social Display Rules Task (SDR) Score | Baseline, 21 weeks
  The SDR task presents 20 hypothetical social scenarios, and asks participants how they should respond to the scenario on a scale ranging from negative to positive responses with 0, 1, or 2 points awarded depending on the response. The test is used to evaluate knowledge of emotional social norms, and scores range from 0 to 40.

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales 21 (DASS-21) Anxiety Scale | Baseline, 21 weeks
  Anxiety symptom severity will be measured with change in the anxiety subscale of the Depression Anxiety Stress Scale-21 (DASS-21). The DASS-21 consists of three 7-item subscales. Participants indicate how much each of 21 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Higher scores indicate higher levels of anxiety.
Change in Depression Anxiety Stress Scales 21 (DASS-21) Stress Scale | Baseline, 21 weeks
  Perceived stress severity will be measured with change in the stress subscale of the Depression Anxiety Stress Scale-21 (DASS-21). The DASS-21 consists of three 7-item subscales. Participants indicate how much each of 21 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Higher scores indicate higher levels of perceived stress.
Change in Depression Anxiety Stress Scales 21 (DASS-21) Depression Scale | Baseline, 21 weeks
  The primary outcome of depression symptom severity will be measured with change in the depression subscale of the Depression Anxiety Stress Scale-21 (DASS-21). The DASS-21 consists of three 7-item subscales. Participants indicate how much each of 21 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Higher scores indicate higher levels of depression.
Change in Difficulties in Emotion Regulation Scale (DERS): Non-acceptance Subscale | Baseline, 21 weeks
  The Difficulties in Emotion Regulation (DERS) test was designed to assess participant's trait-level emotion regulation ability. Responses are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The non-acceptance sub-scale assesses nonacceptance of emotional responses. Scores range from 6 to 30, and higher values reflect greater difficulty with the measured domain.
Change in Difficulties in Emotion Regulation Scale (DERS): Goals Subscale | Baseline, 21 weeks
  The Difficulties in Emotion Regulation-Short Form (DERS) test was designed to assess participant's trait-level emotion regulation ability. Responses are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The goals subscale assesses difficulty engaging in goal-directed behavior. Scores range from 6 to 30, and higher values reflect greater difficulty with the measured domain.
Change in Difficulties in Emotion Regulation Scale (DERS): Impulse Subscale | Baseline, 21 weeks
  The Difficulties in Emotion Regulation (DERS) test was designed to assess participant's trait-level emotion regulation ability. Responses are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The impulse subscale assesses impulse control difficulties. Scores range from 6 to 30, and higher values reflect greater difficulty with the measured domain.
Change in Difficulties in Emotion Regulation Scale (DERS): Awareness Subscale | Baseline, 21 weeks
  The Difficulties in Emotion Regulation (DERS) test was designed to assess participant's trait-level emotion regulation ability. Responses are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The awareness subscale assesses lack of emotional awareness. Scores range from 6 to 30, and higher values reflect greater difficulty with the measured domain.
Change in Difficulties in Emotion Regulation Scale (DERS): Strategies Subscale | Baseline, 21 weeks
  The Difficulties in Emotion Regulation (DERS) test was designed to assess participant's trait-level emotion regulation ability. Responses are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The strategies subscale assesses limited access to emotion regulation strategies. Scores range from 6 to 30, and higher values reflect greater difficulty with the measured domain.
Change in Difficulties in Emotion Regulation Scale (DERS): Clarity Subscale | Baseline, 21 weeks
  The Difficulties in Emotion Regulation (DERS) test was designed to assess participant's trait-level emotion regulation ability. Responses are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The clarity subscale assesses lack of emotional clarity. Scores range from 6 to 30, and higher values reflect greater difficulty with the measured domain.
Change in Scale of Positive and Negative Experiences (SPANE) PA Subscale Score | Baseline, 21 weeks
  The Scale of Positive and Negative Experiences is 12-item self-report measure that will be used to measure a component of subjective well-being, one's positive affect. The subscale ranges from 6 to 30. Higher scores indicate greater experiences of positive affect states (i.e., higher scores on the SPANE-PA scale indicates greater frequency of experiencing positive emotions).
Change in Caregiver Self-Efficacy Score | Baseline, 21 weeks
  A novel 4-item measure on a 1-5 ordinal scale to measure self-efficacy around dementia caregiving. Higher scores represent greater self-efficacy.
Change in Five Facets Mindfulness Questionnaire (FFMQ) Score | Baseline, 21 weeks
  The FFMQ is a 15-item self-reported, instrument assessing mindfulness based on five factors that represent elements of mindfulness ( observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience). Possible scores range from 1 (never or very rarely true) to 5 (very often or always true).
Change in Fears of Compassion Scale (FCS): Fear of Compassion for Self Subscale | Baseline, 21 weeks
  This scale is comprised of 15 items and assesses the compassion we have for ourselves when we make mistakes or things go wrong in our lives. Scores range from 0 to 60. Higher scores indicate greater fear of compassion for self.
Change in Self Compassion Scale Short Form (SCS-SF) Score | Baseline, 21 weeks
  Self Compassion Scale Short Form (SCS-SF) total score, a 12-item self-report measure of self-compassion. The test answers on a Likert scale from 1 to 5, and scores range 12-60 with higher scores indicating greater self compassion.
Change in Hedonic and Eudaimonic Motives for Activities Revised (HEMA-R) Scale | Baseline, 21 weeks
  The HEMA scale is a 10-item questionnaire assessing the extent to which someone values happiness and pleasure versus seeking self-growth, and is measured on a 7-point Likert scale from "not at all" to "very much" for a composite score ranging from 7 to 70. Higher scores indicate better perceived psychological wellbeing.
Change in WHO Quality of Life BREF (WHOQOL BREF) Score | Baseline, 21 weeks
  WHOQOL BREF questionnaire consists of 26 items exploring physical health (7 items), psychological health (6 items), social relations (3 items), environment (8 items) and the quality of life related to health attesting to the overall satisfaction (2 items). Subject responses are collected using a Likert scale, scored from 1 to 5, summed and converted to a scale of 0 (poor quality of life) to 100 (good quality of life). Higher scores indicate better personal quality of life.

OTHER OUTCOMES:
Change in Pleasant Events Schedule (PES-AD) Score | Baseline, 21 weeks
  The Pleasant Events Schedule (PES) will be used to measure the frequency with which the patient engages in enjoyable events. For each of 20 events, caregivers denote the frequency (0 = not at all, 1 = 1-6 times, 2 = 7+ times) with which the patient engaged in the event, and whether the patient enjoyed the event. Higher scores indicate higher frequency and pleasantness of activities.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine P Rankin, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Garland EL, Farb NA, Goldin P, Fredrickson BL. Mindfulness Broadens Awareness and Builds Eudaimonic Meaning: A Process Model of Mindful Positive Emotion Regulation. Psychol Inq. 2015 Oct 1;26(4):293-314. doi: 10.1080/1047840X.2015.1064294. Epub 2015 Nov 24. PMID 27087765
- [Background] Lindsay EK, Creswell JD. Mechanisms of mindfulness training: Monitor and Acceptance Theory (MAT). Clin Psychol Rev. 2017 Feb;51:48-59. doi: 10.1016/j.cpr.2016.10.011. Epub 2016 Nov 5. PMID 27835764
- [Background] Li G, Yuan H, Zhang W. The Effects of Mindfulness-Based Stress Reduction for Family Caregivers: Systematic Review. Arch Psychiatr Nurs. 2016 Apr;30(2):292-9. doi: 10.1016/j.apnu.2015.08.014. Epub 2015 Aug 28. PMID 26992885
- [Background] Steadman PL, Tremont G, Davis JD. Premorbid relationship satisfaction and caregiver burden in dementia caregivers. J Geriatr Psychiatry Neurol. 2007 Jun;20(2):115-9. doi: 10.1177/0891988706298624. PMID 17548782
- [Background] Campos D, Modrego-Alarcon M, Lopez-Del-Hoyo Y, Gonzalez-Panzano M, Van Gordon W, Shonin E, Navarro-Gil M, Garcia-Campayo J. Exploring the Role of Meditation and Dispositional Mindfulness on Social Cognition Domains: A Controlled Study. Front Psychol. 2019 Apr 11;10:809. doi: 10.3389/fpsyg.2019.00809. eCollection 2019. PMID 31031678
- [Background] Luberto CM, Shinday N, Song R, Philpotts LL, Park ER, Fricchione GL, Yeh GY. A Systematic Review and Meta-analysis of the Effects of Meditation on Empathy, Compassion, and Prosocial Behaviors. Mindfulness (N Y). 2018 Jun;9(3):708-724. doi: 10.1007/s12671-017-0841-8. Epub 2017 Oct 23. PMID 30100929